CLINICAL TRIAL: NCT05332938
Title: Impact of Acetabular Fractures on Sports Performance
Acronym: Fracture&Sport
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Fracture&Sport
Record Dates: First submitted 2022-04-01; First posted 2022-04-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetabular fractures are complex, relatively rare lesions that are difficult to manage. Given the surgical challenge they represent, they are often managed by expert centers. The overall incidence of these fractures is around 3 fractures/100,000 persons/year.

It is now well established that the quality of the reduction obtained is an important predictive factor of the postoperative outcome in patients with displaced acetabular fractures. Obtaining an anatomical reduction, at least satisfactory, is not always easy, even in trained teams. Indeed, it can be difficult because of the structural environment. This is due to the proximity of the acetabulum to the vasculo-nervous elements, but also to the complexity of the fracture itself. The contribution of new technologies appear to be important tools to achieve this objective. Indeed, investigators have demonstrated that the use of the O-ARM imaging system (Medtronic®, Sofamor, Memphis, TN) allowed the improvement of their results.

Although they occur more frequently in the elderly population, the average incidence is maintained in the 20-59 age group. In these young populations, the fracture occurs most frequently as a result of a high-energy mechanism (road accident, more exceptionally, during a sporting activity). These patients, in the prime of their lives, are often athletic. The desire to resume sports after surgery is a powerful motivating factor for these patients. Often, it is the primary measure of surgical success from the athlete's perspective. In a previous work, Giannoudis et al. reported a 42% rate of return to activity at the previous level. The quality of the surgery is associated with the possibility of resuming sports activity after the procedure.

Thus, the objective of this work is to determine the results of acetabular surgery in a population of previously athletic patients, in particular the return to athletic performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 45 years at the time of surgery at Saint Joseph Hospital
* Patients with an isolated acetabulum fracture
* Patients with intraoperative management with O-Arm
* Patients with at least 2 years of follow-up
* French-speaking patients

Exclusion Criteria:

* Presence of pre- or post-operative neurological lesions
* Presence of associated fractures
* ASA (American Society of Anesthesiologists) score ≥ 3
* Absence of pre- and postoperative CT scans available on PACS
* Patients under guardianship or curatorship
* Patients deprived of liberty
* Patients under court protection
* Patients objecting to participation in the study
* Low preoperative physical activity (= UCLA Activity Score ≤ 5)
* Unsatisfactory criteria for surgical reduction on CT scan

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients aged 18 to 45 years at the time of surgery at Saint Joseph Hospital, victims of an isolated acetabulum fracture, having received intraoperative management with O-ARM, with at least 2 years of follow-up
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients returning to sports after surgery at 2 years | Year 2
  This outcome corresponds to the number of patients who have returned to sport at the same level, performing at or above their pre-injury level, without time limitation.

SECONDARY OUTCOMES:
Complication rate | Year 2
  This outcome corresponds to the number of patients with postoperative complications (infection, hematoma, anemia requiring transfusion).
Quality of sports recovery at 2 years | Year 2
  This outcome corresponds to the time to resume performance.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Lundin N, Huttunen TT, Berg HE, Marcano A, Fellander-Tsai L, Enocson A. Increasing incidence of pelvic and acetabular fractures. A nationwide study of 87,308 fractures over a 16-year period in Sweden. Injury. 2021 Jun;52(6):1410-1417. doi: 10.1016/j.injury.2021.03.013. Epub 2021 Mar 14. PMID 33771345
- [Background] Tannast M, Najibi S, Matta JM. Two to twenty-year survivorship of the hip in 810 patients with operatively treated acetabular fractures. J Bone Joint Surg Am. 2012 Sep 5;94(17):1559-67. doi: 10.2106/JBJS.K.00444. PMID 22992846
- [Background] Giannoudis PV, Grotz MR, Papakostidis C, Dinopoulos H. Operative treatment of displaced fractures of the acetabulum. A meta-analysis. J Bone Joint Surg Br. 2005 Jan;87(1):2-9. PMID 15686228
- [Background] Ziran N, Soles GLS, Matta JM. Outcomes after surgical treatment of acetabular fractures: a review. Patient Saf Surg. 2019 Mar 16;13:16. doi: 10.1186/s13037-019-0196-2. eCollection 2019. PMID 30923570
- [Background] Rizkallah M, Sebaaly A, Melhem E, Moreau PE, Upex P, Jouffroy P, Riouallon G. Clinical impact of intraoperative cone beam tomography and navigation for displaced acetabular fractures: a comparative study at medium-term follow-up. Int Orthop. 2021 Jul;45(7):1837-1844. doi: 10.1007/s00264-021-05076-4. Epub 2021 May 22. PMID 34021374
- [Background] Melhem E, Riouallon G, Habboubi K, Gabbas M, Jouffroy P. Epidemiology of pelvic and acetabular fractures in France. Orthop Traumatol Surg Res. 2020 Sep;106(5):831-839. doi: 10.1016/j.otsr.2019.11.019. Epub 2020 Feb 1. PMID 32019733
- [Background] Doege J, Ayres JM, Mackay MJ, Tarakemeh A, Brown SM, Vopat BG, Mulcahey MK. Defining Return to Sport: A Systematic Review. Orthop J Sports Med. 2021 Jul 26;9(7):23259671211009589. doi: 10.1177/23259671211009589. eCollection 2021 Jul. PMID 34377709
- See also: Related Info — https://www.researchgate.net/publication/352127142_Computed_tomography_assessment_of_low-energy_acetabular_fractures_in_the_elderly